CLINICAL TRIAL: NCT07019896
Title: Minimal Vitrectomy Surgery (MVS) Versus Conventional Vitrectomy for the Treatment of Idiopathic Epiretinal Membrane: A Multicenter Randomized Controlled Trial
Brief Title: Minimal Vitrectomy Surgery for Epiretinal Membrane
Acronym: MVS-ERM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Weihong Yu, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-I2M-C&T-B-028; K4698 (Other: Peking Union Medical College Hospital)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Epiretinal Membrane; Macular Edema (ME); Nuclear Cataract
Keywords: Idiopathic Epiretinal Membrane (ERM); Minimal Vitrectomy Surgery (MVS); Nonvitrectomizing Vitreous Surgery (NVS); pars plana Vitrectomy (PPV)
MeSH Terms: conditions — Epiretinal Membrane; Macular Edema

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, randomized, parallel-group controlled trial. Patients with idiopathic epiretinal membrane are randomly assigned to receive either Minimal Vitrectomy Surgery (MVS) or Conventional Pars Plana Vitrectomy (PPV). Randomization is stratified across 14 participating centers. Participants in the MVS group undergo membrane peeling without core vitrectomy or posterior vitreous detachment induction, with selective limited vitrectomy performed if necessary. The PPV group undergoes standard vitrectomy with core vitreous removal and posterior vitreous detachment prior to membrane peeling.
Who Masked: Participant
Masking Description: Participants are masked to the intervention arm assignment. Surgical staff, investigators, and outcomes assessors are not masked due to the nature of the surgical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Vitrectomy Surgery (MVS) (Experimental): The epiretinal membrane is peeled directly through the intact vitreous. Limited vitrectomy is selectively performed if pre-existing floaters or membrane fragments remain after peeling and cannot be removed safely with forceps.
  Interventions: Procedure: Minimal Vitrectomy Surgery
- Conventional Vitrectomy (PPV) (Active Comparator): Standard pars plana vitrectomy is performed. Posterior vitreous detachment induction and core vitreous removal are conducted before membrane peeling.
  Interventions: Procedure: Conventional Vitrectomy

INTERVENTIONS:
Procedure: Minimal Vitrectomy Surgery — The epiretinal membrane is peeled directly through the intact vitreous. Limited localized vitrectomy is selectively performed if pre-existing floaters or membrane fragments remain after peeling.
  Arms: Minimal Vitrectomy Surgery (MVS)
Procedure: Conventional Vitrectomy — Standard pars plana vitrectomy is performed with posterior vitreous detachment induction and core vitreous removal prior to epiretinal membrane peeling.
  Arms: Conventional Vitrectomy (PPV)

SUMMARY:
This multicenter randomized controlled trial evaluates Minimal Vitrectomy Surgery (MVS) versus conventional vitrectomy for idiopathic epiretinal membrane (ERM). The primary endpoints include visual acuity improvement and cataract progression after 12 months. MVS aims to minimize vitreous removal while ensuring complete membrane removal through adaptive limited vitrectomy.

DETAILED DESCRIPTION:
Idiopathic epiretinal membrane (ERM) is characterized by fibrocellular proliferation on the retinal surface, leading to macular edema, metamorphopsia, and visual impairment. Traditional treatment involves pars plana vitrectomy (PPV) with posterior vitreous detachment (PVD) induction and core vitrectomy, which may increase the risk of postoperative cataract.

Minimal Vitrectomy Surgery (MVS) is a modified surgical approach designed to minimize vitreous removal and preserve the hyaloid. The epiretinal membrane is directly peeled through the intact vitreous. If pre-existing vitreous floaters or membrane fragments remain after peeling and cannot be removed safely with micro-forceps, limited localized vitrectomy is selectively performed to eliminate these floaters and avoid postoperative visual disturbances.

This trial aims to evaluate the efficacy and safety of MVS compared to conventional vitrectomy, focusing on visual improvement, macular thickness, cataract progression, ERM recurrence, and intraoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosis of idiopathic epiretinal membrane (ERM) confirmed by clinical examination and OCT imaging.
3. Clear ocular media allowing adequate fundus imaging.
4. Phakic eye.
5. Ability and willingness to provide written informed consent.

Exclusion Criteria:

1. Prior cataract surgery or advanced cataract requiring combined surgery. Co-existing retinal diseases (e.g., diabetic retinopathy, retinal detachment, retinal vein occlusion).
2. Systemic conditions preventing safe surgery or follow-up.
3. History of prior ocular or periocular corticosteroid use, including intraocular injection, periocular injection, or long-term topical corticosteroid eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Cataract progression assessed by LOCS III and DLI | Baseline, 12 months
  Cataract progression evaluated by Lens Opacities Classification System III (LOCS III) grading and Dysfunctional Lens Index (DLI) changes.

SECONDARY OUTCOMES:
BCVA change from baseline to 12 months | Baseline, 1 week, 1 month, 3 months, 6 months, 12 months
  Change in best-corrected visual acuity (logMAR) from baseline to 12 months postoperatively.
Change in central retinal thickness (CRT) by OCT | Baseline, 1 week, 1 month, 3 months, 6 months, 12 months
  Change in macular central retinal thickness as assessed by OCT.
Epiretinal membrane recurrence rate | 12 months
  Recurrence of epiretinal membrane at 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Weihong Yu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient privacy protection and the absence of participant consent for data sharing. The study data will be used exclusively for internal research purposes and regulatory submissions.